CLINICAL TRIAL: NCT02104414
Title: Comparison of Rectal Infiltration of Exparel vs. 0.25% Bupivacaine With Epinephrine vs. Placebo for Analgesic Benefit Following Hemorrhoidectomy
Brief Title: Efficacy of Rectal Infiltration of Exparel for Analgesic Benefit Following Hemorrhoidectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-0062
Record Dates: First submitted 2014-03-28; First posted 2014-04-04 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Hemorrhoid
Keywords: Liposomal Bupivacaine; Exparel
MeSH Terms: conditions — Hemorrhoids | interventions — Bupivacaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Exparel (Active Comparator): 266mg/20mL Exparel (to be diluted with 10 mL sterile saline to make 30 mL)
  Interventions: Drug: Exparel
- Bupivacaine HCl with epinephrine (Active Comparator): 75mg/30mL 0.25% Bupivacaine HCl with epinephrine
  Interventions: Drug: Bupivacaine HCl with Epinephrine
- Normal Saline (Placebo Comparator): 30mL Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Exparel — 266 mg/20mL Exparel (to be diluted with 10 mL sterile saline to make 30 mL)
  Other Names: Liposomal Bupivacaine
  Arms: Exparel
Drug: Bupivacaine HCl with Epinephrine — 75mg/30mL 0.25% Bupivacaine HCl with epinephrine
  Arms: Bupivacaine HCl with epinephrine
Drug: Normal Saline — 30mL Normal Saline
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to compare the quality and duration of pain relief after a hemorrhoidectomy, provided by locally administered liposomal bupivacaine versus bupivacaine hcl or control with saline. It is hypothesized that liposomal bupivacaine will provide more effective postoperative pain relief than both bupivacaine hcl and the control.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hemorrhoidectomy for grade 3 or 4 hemorrhoids who are English-speaking patients, 21-65 yr of age, ASA physical status I-III, BMI<30

Exclusion Criteria:

* contraindications to administration of local anesthesia (e.g., local anesthetic allergy), difficult airway (Mallampati>2), psychiatric or cognitive disorders, pregnancy , and history of substance abuse or chronic opioid use

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shariat, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St.Luke's-Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Started | 5 | 4 | 2
Completed | 5 | 4 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline | Total
Number analyzed (Participants) | 5 | 4 | 2 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (14.61) | 40.75 (13.1) | 51.5 (9.19) | 44.54 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 4 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain Control
Description: The primary objective is to evaluate analgesia following local infiltration of 30 mL Exparel or the same volume of 0.25% bupivacaine HCl with epinephrine or normal saline. The intensity of pain will be measured using a numerical rating scale (NRS-11) in which 0 represents no pain, and 10 represents extreme pain.
Time Frame: up to 4 days
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
score on a scale
  Hour 1 | 0 [0 to 10] | 1.33 [0 to 10] | 7 [0 to 10]
  Hour 2 | 0 [0 to 10] | 1.0 [0 to 10] | 2.5 [0 to 10]
  Day 1 | 5.75 [0 to 10] | 6.5 [0 to 10] | 5.5 [0 to 10]
  Day 2 | 3 [0 to 10] | 4.5 [0 to 10] | 4 [0 to 10]
  Day 3 | 2.25 [0 to 10] | 5.0 [0 to 10] | 3 [0 to 10]
  Day 4 | 2.67 [0 to 10] | 3.0 [0 to 10] | 2 [0 to 10]

2. Secondary Outcome: Number of Oxycodone Tablets Taken
Description: Number of postoperative opioid consumption - oxycodone tablets (5mg each)
Time Frame: up to 4 days
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
tablets
  Hour 1 | 0 (0) | 0 (0) | 0 (0)
  Hour 2 | 0 (0) | 0 (0) | 0 (0)
  Day 1 | 2.2 (2.28) | 2.67 (1.53) | 1.5 (0.71)
  Day 2 | 2 (1.58) | 1.67 (0.58) | 2.5 (0.71)
  Day 3 | 1.4 (1.52) | 1.5 (0.78) | 2.5 (0.71)
  Day 4 | 2 (1.63) | 1 (0) | 1.5 (0.71)

3. Secondary Outcome: Postoperative Opioid Consumption - Hydromorphone I.V
Time Frame: 1 hour and 2 hours post op
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
mg
  Hour 1 | 0.35 (0.47) | 0 (0) | 0.8 (0.42)
  Hour 2 | 0.5 (0.6) | 0 (0) | 0.6 (0.28)

4. Secondary Outcome: Number of Participants With Postoperative Nausea and Vomiting
Description: Number of participants with postoperative nausea and vomiting episodes
Time Frame: up to 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
Participants
  Hour 1 | 0 | 0 | 0
  Hour 2 | 0 | 0 | 0
  Day 1 | 0 | 0 | 0
  Day 2 | 0 | 0 | 0
  Day 3 | 0 | 0 | 0
  Day 4 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Pain During Bowel Movements
Description: Number of participants with pain during postoperative bowel movements
Time Frame: Hourly from PACU arrival to discharge and Q4H from 10:00-22:00 postoperatively for 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
Participants
  Day 1 | 1 | 1 | 1
  Day 2 | 2 | 3 | 1
  Day 3 | 5 | 4 | 2
  Day 4 | 5 | 4 | 2

6. Secondary Outcome: Number of Participants With Urinary Retention
Time Frame: up to 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
Number analyzed (Participants) | 5 | 4 | 2
Participants
  Day 1 | 0 | 0 | 0
  Day 2 | 0 | 0 | 0
  Day 3 | 0 | 0 | 0
  Day 4 | 0 | 0 | 0

ADVERSE EVENTS:
Description: There were no adverse events
Arm/Group | Exparel | Bupivacaine HCl With Epinephrine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes